CLINICAL TRIAL: NCT06901375
Title: 14-day Zuojin Wan Combined with Vonoprazan-Amoxicillin Dual Therapy in the Treatment of Helicobacter Pylori Associated Chronic Gastritis:A Single-Center,Randomized Controlled Study
Brief Title: Zuojin Wan Combined with Vonoprazan-Amoxicillin Dual Therapy in H.Pylori Eradication
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20240613-11-KS-01
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-06

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; zuojin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonoprazan-amoxicillin dual therapy (Active Comparator): Participants received Vonoprazan 20 mg tablet orally twice daily and Amoxicillin 1 g tablet orally three times daily for 2 weeks.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- Zuojin Wan ombined with vonoprazan-amoxicillin dual therapy (Experimental): Participants received Vonoprazan 20 mg tablet,Zuojin Wan 3 g tablet orally twice daily and Amoxicillin 1 g tablet orally three times daily for 10 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Zuojin Wan

INTERVENTIONS:
Drug: Vonoprazan — 20 mg tablet twice daily
  Other Names: Vonoprazan fumarate
Drug: Amoxicillin — 1 g tablet three times daily
  Other Names: Amoxicillin Capsules
Drug: Zuojin Wan — 3 g tablet twice daily
  Other Names: Zuojin Pill
  Arms: Zuojin Wan ombined with vonoprazan-amoxicillin dual therapy

SUMMARY:
Vonoprazan and high-dose amoxicillin dual therapy was used as a control group to evaluate the clinical efficiency and safety of Zuojin Wan combined with vonoprazan and high-dose amoxicillin dual therapy in the treatment of helicobacter pylori associated chronic gastritis,through a randomized controlled trail.

DETAILED DESCRIPTION:
Helicobacter pylori（H.pylori）is a gastric pathogen, related to various gastrointestinal disorders. It's now a consensus of experts that H.pylori infection should be treated once it is recognized. Vonoprazan and high-dose amoxicillin dual therapy is a potential H.pylori eradication regimen. It provides a satisfactory eradication rate of 90%. Nevertheless,it has certain limitations, including a series of problems such as low eradication rate and more side effects of eradication in recurrent patients. The main side effects of the dual therapy for eradication are related symptoms of gastric motility deficiency and indigestion, such as bloating, abdominal pain, belching, acid reflux, etc. Combining traditional Chinese medicine may be one of the effective ways to solve the above problems.This study aims to compare the efficacy of Zuojin Wan combined with vonoprazan and high-dose amoxicillin dual therapy,with that of vonoprazan and high-dose amoxicillin dual therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Patients with H.pylori infection
3. Diagnosed as functional dyspepsia
4. Meet the diagnostic criteria of H. pylori liver-atomach stagnation heat syndrome in traditional Chinese medicine.
5. Patients who have not received H. pylori eradication treatment before, or who have failed eradication in the early stage but have not received eradication treatment within six months.
6. Volunteer to participate in this experiment and sign the informed consent.

Exclusion Criteria:

1. Allergy to research drugs (penicillin allergy, etc.)
2. Patients with gastric and duodenal ulcer, pyloric obstruction, esophageal and gastric varices, gastrorrhagia, gastrointestinal mucosa with dysplasia, gastric malignant tumor and other gastrointestinal diseases.
3. Patients with severe heart, brain, liver, kidney, hematopoietic system and connective tissue diseases
4. Patients who have received H. pylori eradication treatment within six months.
5. Antibiotics and bismuth were used 4 weeks before the start of study treatment, and histamine H2 receptor antagonist or PPI was used 2 weeks before the start of study treatment.
6. Use adrenocortical hormone, non-steroidal anti-inflammatory drugs or anticoagulants.
7. History of esophageal or gastric surgery
8. Pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in functional dyspepsia symptoms at 6 weeks | Baseline and Week 6
  Dyspepsia symptoms on days 7,14 and 42 were assessed using Likert scale； Scale tittle:Symptom frequency and severity criteria table； The minimum value：8；the maximum value：40； Higher scores mean a worse outcome.
Change in Traditional Chinese Medicine syndromes from Baseline to 6 weeks | Baseline and Week 6
  Traditional Chinese Medicine syndromes on days 7,14 and 42 were assessed using Traditional Chinese Medicine syndrome integral scale.Scale tittle:Traditional Chinese Medicine syndrome integral scale; The minimum value：0；the maximum value：30； Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Adverse events during the treatment | day 1 and day 14
  The occurrence of adverse events during treatment will be recorded by telephone follow-up.
Patients' drug compliance | day 1 and day 14
  Patients' drug compliance was assessed using medication possession ratio

CONTACTS AND LOCATIONS:
Overall Officials: Wanli Liu, Doctorate, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospitai, Nanjing, Jiangsu, China